CLINICAL TRIAL: NCT05717010
Title: Is There a Risk of Perioperative Stroke Due to the Retraction Used During Anterior Cervical Discectomy?
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: Samsun University (SamsunU)
Record Dates: First submitted 2022-12-16; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Cervical Disc Disease; Cervical Stenosis; Cervical Disc Herniation
Keywords: Cerebral blood oxygenation; Near infrared spectroscopy; Cervical disc disease; Cervical microsurgery
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days

GROUPS / COHORTS (2):
- Group self-retaining retractor: Patients used self-retaining retractor for surgery
  Interventions: Device: Near infrared spectroscopy
- Group Hand-held retractor: Patients used hand held retractor for surgery
  Interventions: Device: Near infrared spectroscopy

INTERVENTIONS:
Device: Near infrared spectroscopy — The Near Infrared Spectroscopy (NIRS) is the method used for monitorize the risk of the development of cerebral ischaemia while providing information about brain tissue oxygenation.

SUMMARY:
In anterior cervical disc surgery, head and neck extansion position and, surgical retraction used while reaching the anterior surface of the cervical vertebra can be affect the carotid blood flow and constituting a risk for cerebral ischaemia. In this study, we planned to investigate the relationship between head position and retraction, cerebral oxygenation and postoperative cognitive functions in patients undergoing anterior cervical disc surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years
* Preoperative Mini-Mental State Examination score of 27-30
* Who were planned to undergo anterior cervical disc surgery under general anesthesia

Exclusion Criteria:

* Patients with hypertension, severe pulmonary disease, anaemia, cardiac disease, ischaemic cerebrovascular disease, renal disease, hepatic disease, pregnancy, uncontrolled diabetes mellitus, stricture or obstruction in the carotid or vertebral arteries or
* Body mass index (BMI) >30.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cervical disc surgery
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Near-infrared spectroscopy (NIRS) | Intraoperative
  Evaluate the effect of head position and surgical retraction on brain oxygenization with NIRS. Near-infrared spectroscopy (NIRS) is a brain imaging method that measures light absorbance to calculate oxy-hemoglobin (oxy-HB) and deoxy-hemoglobin (deoxy-HB), which provides an indirect measure of brain activity, particularly in the frontal cortex.

SECONDARY OUTCOMES:
Mini-Mental State Examination | 2 hours postoperative
  Evaluate the effect of head position and surgical retraction on cognitive functions with using mini-mental state examination . A Mini-Mental State Examination (MMSE) is a set of 30 questions that commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory)

CONTACTS AND LOCATIONS:
Overall Officials: Samsun Üniversitesi, Study Chair — Samsun University
Locations (1):
- Nevin Esra Gumus, Samsun, Turkey (Türkiye)

REFERENCES:
- [Result] Smarius BJA, Breugem CC, Boasson MP, Alikhil S, van Norden J, van der Molen ABM, de Graaff JC. Effect of hyperextension of the neck (rose position) on cerebral blood oxygenation in patients who underwent cleft palate reconstructive surgery: prospective cohort study using near-infrared spectroscopy. Clin Oral Investig. 2020 Aug;24(8):2909-2918. doi: 10.1007/s00784-019-03157-8. Epub 2020 Mar 26. PMID 32219565